CLINICAL TRIAL: NCT01631110
Title: Open, Non-randomized Trial to Assess the Immunogenicity and Safety of the 2012/2013-Season Influenza Vaccine in Elderly and Young Subjects According to EMA Regulations
Brief Title: Re-licensing Study to Assess Inflexal V Formulated With WHO Recommended Influenza Strains
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INF-V-A010
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Inflexal V
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Inflexal V; Antigens, Surface; Virosomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly subjects aged over 60 years (Experimental)
  Interventions: Biological: Inflexal V
- Adults from 18 to 60 years old inclusive (Experimental)
  Interventions: Biological: Inflexal V

INTERVENTIONS:
Biological: Inflexal V — Intramuscular administration (M. deltoideus) of a single dose of 0.5 mL Inflexal V
  Other Names: Inflexal V influenza vaccine (surface antigen, inactivated, virosome) formulated for the WHO requirements of the 2012-2013 season, each 0.5 mL dose containing:; • 15 µg HA antigen of A/California/7/2009 (H1N1)-like virus; • 15 µg HA antigen of A/Victoria/361/2011 (H3N2)-like virus; • 15 µg HA antigen of B/Wisconsin/1/2010-like virus

SUMMARY:
The study is to assess whether the influenza vaccine Inflexal V for season 2012/2013 fulfills the EMA requirements for re-registration of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults aged ≥18 on Day 1
* Written informed consent
* Female subjects of childbearing potential using and willing to continue using an acceptable method of contraception unless surgically sterilized/hysterectomized or post-menopausal for more than 2 years

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine in the past 330 days
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, including oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (incl. leukemia, HIV seropositivity), cancer
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial
* Employee at the investigational site, or relative of the investigator
* Subjects who in the view of the investigator will not comply with study procedures and/or visit requirements as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — Covance Clinical Research Unit AG
Locations (1):
- Covance Clinical Research Unit AG, Allschwil, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 23 July 2012 to 14 August 2012; outpatient study
Period: Overall Study
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 55 | 78
  >=65 years | 32 | 0 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (6.01) | 38.3 (11.69) | 52.8 (17.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 33 | 31 | 64
Region of Enrollment [Number; unit: participants]
  Switzerland | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection
Description: Seroprotection rate, defined as proportion of subjects with HI antibody titer ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: Day 22 +/- 2 days
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
percentage of subjects
  Percentage seroprotected subjects: A/H1N1 | 65.5 [51.4 to 77.8] | 80.0 [67.0 to 89.6]
  Percentage seroprotected subjects: A/H3N2 | 98.2 [90.3 to 100] | 98.2 [90.3 to 100]
  Percentage seroprotected subjects: B strain | 52.7 [38.8 to 66.3] | 70.9 [57.1 to 82.4]

2. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events, as a Measure of Safety and Tolerability
Description: Solicited local and systemic AEs, Unsolicited AEs
  Unsolicited AEs were collected from baseline (Day 1) to 3 weeks after vaccination (Day 22 ± 2 days).
  Solicited local and systemic AEs were collected by subjects diary from Day 1 (day of vaccination) to Day 4
Time Frame: Baseline (Day 1) and 3 weeks after vaccination (Day 22 ± 2 days)
Population: Safety population, all vaccinated subjects
Measure: Number; unit: Participants
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
Participants
  AEs (unsolicited and unsolicited) | 25 | 35
  Unsolicited AEs | 10 | 10
  Solicited local AEs | 17 | 33
  Solicited systemic AEs | 3 | 2

3. Primary Outcome: Seroconversion
Description: Seroconversion rate, defined as proportion of subjects with ≥4-fold increase in HI antibody titer and with a titer of ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: Day 22 +/- 2 days
Population: Intent-to-treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
percentage of subjects
  Percentage seroconverted subjects: A/H1N1 | 50.9 [37.1 to 64.6] | 45.5 [32.0 to 59.4]
  Percentage seroconverted subjects: A/H3N2 | 18.2 [9.1 to 30.9] | 12.7 [5.3 to 24.5]
  Percentage seroconverted subjects: B strain | 25.5 [14.7 to 39.0] | 41.8 [28.7 to 55.9]

4. Primary Outcome: Geometric Mean Titer
Description: GMT of HI antibodies and fold-increase in GMT (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: Day 22 +/- 2 days
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: GMT fold increase from baseline
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
GMT fold increase from baseline
  GMT fold increase: A/H1N1 | 5.15 [3.55 to 7.45] | 4.36 [3.32 to 5.71]
  GMT fold increase: A/H3N2 | 1.96 [1.64 to 2.35] | 1.72 [1.49 to 1.99]
  GMT fold increase: B strain | 2.40 [1.97 to 2.92] | 3.33 [2.55 to 4.36]

ADVERSE EVENTS:
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 25/55 | 35/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderly Subjects Aged Over 60 Years (N=55) | Adults From 18 to 60 Years Old Inclusive (N=55)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Vessel puncture swelling (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 6 (6) | 7 (7)
Injection site haemorrhage (General disorders) | 2 (2) | 4 (4)
Injection site induration (General disorders) | 3 (3) | 6 (6)
Injection site pain (General disorders) | 10 (10) | 27 (27)
Malaise (General disorders) | 2 (2) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 7 (7)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Material for public dissemination will be submitted to the sponsor for review at least ninety (90) days prior to submission for publication, public dissemination, or review by a publication committee.